CLINICAL TRIAL: NCT03671941
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate Pharmacokinetic Profiles and Safety/Tolerability of CKD-357 in Healthy Volunteers
Brief Title: Clinical Study to Compare the Pharmacokinetic Characteristics and Safety Between CKD-357 and D578 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 180BE18003
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): D578 Tab. 1T
  Interventions: Drug: D578
- Group B (Experimental): CKD-357 Tab. 1T
  Interventions: Drug: CKD-357

INTERVENTIONS:
Drug: D578 — D578 Tab.1T single oral administration under fasting condition
  Other Names: Ticagrelor
  Arms: Group A
Drug: CKD-357 — CKD-357 Tab.1T single oral administration under fasting condition
  Other Names: Novel salts of Ticagrelor
  Arms: Group B

SUMMARY:
A randomized, open-label, single dose, crossover study to evaluate pharmacokinetic profiles and safety/tolerability of CKD-357 in healthy volunteers

DETAILED DESCRIPTION:
To healthy subjects of thirty(30), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

ELIGIBILITY:
[Inclusion Criteria]

1. A healthy adult whose age is over 19 years old when visiting for initial screening test
2. Body mass index(BMI) between 17.5~30.5 kg/m^2 and the body weight must be over 55kg (Body mass index (BMI) = weight (kg) / height (m)^2)
3. A person with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening after examined through hematology test and blood chemistry analysis, urinary test, viral/bacterial test, the electrocardiogram (ECG), and etc.
5. The participants must be volunteered and sign in an informed consent document proven by Chonbuk National University IRB before joining a study to show that he was given informed the purpose of tests and the special characteristics of drugs.
6. The participants must have an ability and willingness to participate throughout the entire trials

[Exclusion Criteria]

1. A person who had a history or symptoms of clinically aware of blood, kidney, internal secretion, respiratory, gastrointestinal, urinary system, cardiovascular, liver, mental, nervous, or allergic(except subclinical seasonal allergies that is not treated at injection) disease.
2. Who had a history of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy)
3. Who had following results after examination

   a. ALT or AST > twice higher than normal value
4. Who constantly intake 210 g/week of alcohol within 6 months of the screening. (a cup of beer (5%) (250 mL) = 10 g, a shot of soju (20%) (50mL) = 8 g, a glass of wine (!2%) (125 mL) = 12g)
5. Who participated other clinical test or took testing bioequivalence drugs in 3 months before the first clinical drug trial.
6. Whose blood pressure < 100 or ≥140(systolic blood pressure) or < 70 or ≥ 90(diastolic blood pressure)
7. Who had a medical history of alcohol and drug abuses.
8. Who had taken a drug that has a control of metabolic rate (activation or inhibition) in 30 days before the first taking of clinical testing durg.
9. Who smokes more than 20 cigarettes per day within 6 months of the screening
10. Who took prescribed drugs or over-the-counter drugs in 10 days before taking of very first clinical testing drug.
11. Who participated in whole blood donation in 2 months before the first taking of clinical testing drugs or platelet donations in 1 month before the first taking to clinical testing drugs
12. Who has a potent to increase a danger by participating in the clinical trials or sho can interrupt interpreting test results by having serious or chronic medical and mental status or having issues in results of the screening examination.
13. Who has a history of an extreme sensitivity of composition of the drug
14. Who has hemorrhagic tendency(recently trauma, recently surgery, coagulation disorder, recently gastrointestinal bleeding)and are scheduled for surgery within one month
15. Who has a potent to increase a danger of beat heart slowly like symptom of bradycardia and dyspnea
16. Who had a medical history of hyperuricacidemia and gouty arthritis
17. Who has a Pregnant or potentially pregnant.
18. A person who is not determined unsuitable to participate in this test by the researchers

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
AUCt of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Area under the plasma concentration of Ticagrelor versus time curve from time zero to time of last quantifiable concentration
Cmax of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Maximum plasma concentration of Ticagrelor

SECONDARY OUTCOMES:
AUCinf of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Area under the plasma concentration of Ticagrelor versus time curve from time zero to time infinity
Tmax of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Time to maximum concentration of of Ticagrelor
t1/2 of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent terminal half-life of Ticagrelor
CL/F of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Total body clearance of Ticagrelor
Vd/F of Ticagrelor | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Apparent volume of distribution of Ticagrelor
AUCt of AR-C124910XX | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Area under the plasma concentration of AR-C124910XX versus time curve from time zero to time of last quantifiable concentration
Cmax of AR-C124910XX | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Maximum plasma concentration of AR-C124910XX
AUCinf of AR-C124910XX | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Area under the plasma concentration of AR-C124910XX versus time curve from time zero to time infinity
Tmax of AR-C124910XX | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Time to maximum concentration of AR-C124910XX
t1/2 of AR-C124910XX | Pre-dose(0 hour), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Apparent terminal half-life of AR-C124910XX

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Ho Jang, Professor, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea